CLINICAL TRIAL: NCT03762733
Title: Tissue Acquisition and Genomics Analysis of Breast Cancer and Other Gynecologic Malignancies
Status: Enrolling by invitation | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 190025; 19-C-0025
Record Dates: First submitted 2018-12-01; First posted 2018-12-04 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01-15

CONDITIONS: Breast Cancer; Ovarian Cancer; Uterine Cancer
Keywords: Biobanking; Tissue Repository; Genetic Analysis; Natural History
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Uterine Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient Relatives: Biological relatives (1st-3rd degree) of participants with histologically confirmed malignancy
- Patients: Participants with histologically confirmed malignancy

SUMMARY:
Background:

A person s blood, tissue, and other samples contain DNA. Cancer is a disease of cells that are not working properly. It is caused by changes in DNA that build up. Researchers want to do future studies on DNA changes This may help them learn how to guide treatment for cancer. They need biological samples like tumors, blood, and urine for these studies.

Objective:

To create a place to collect and store biological samples from people with gynecologic malignancies like breast cancer. Samples from certain relatives of theirs will be collected too.

Eligibility:

Adults ages 18 and older who are being seen at NIH for breast cancer or other gynecologic malignancy

Their biological relatives of the same age

Design:

Participants will answer questions about their family history.

Participants will have a physical exam and medical history. This will include questions about age, ethnicity, and disease history. They will also answer questions about their medical treatments and responses.

Participants will give blood and urine samples.

Participants may give a tumor tissue sample. This will not be taken specifically for this study. It will be from a previous procedure or one that is already planned.

Other samples may be taken only if a procedure is required for treatment. These include bone marrow, cerebrospinal fluid, and other fluids.

A group of doctors and other professionals will oversee the sample storage place. The group will review all requests to be sure the use of the specimens is valid.

DETAILED DESCRIPTION:
Background:

Increased understanding of the genomic variations of cancer through laboratory evaluations can result in breakthroughs in treatment and improved patient outcomes.

Exceptional responders on clinical trials may have mutational characteristics that are unique and unknown, necessitating identification.

Current drug development strategies employ precision oncology. This approach identifies molecular targets, with therapies being either chosen or developed to interact with the specific target.

The collection and banking of a variety of tissue samples for future translational studies would support research and advance the mission of the NIH.

Pleural effusions, ascites as well as other tissues, such as blood, CSF, tumor, bone marrow, and urine, provide a unique opportunity to conduct a variety of translational research, addressing many clinical questions.

The establishment of a tissue repository would enhance the mission of the NCI, in helping to advance research supporting precision oncology.

Primary Objective:

To establish a tissue repository for the collection and banking of tissue samples from patients with breast and/or other gynecologic malignancies, as well as patients consenting 1st -3rd degree biological relatives, seen at the NIH for support of future translational research conducted at the NIH.

Eligibility:

Personal diagnosis of breast or other gynecologic malignancy, or be a 1st-3rd degree biological relative of a patient with cancer, currently or previously on a NIH clinical trial.

All subjects (index patient with cancer and their 1st-3rd degree biological relatives) must sign consent and enroll onto this study, in order to donate tissue for biobanking on this protocol.

Adults, >= age 18, willing to provide tissue for biobanking

Design:

Samples include, but are not limited to, tumor (e.g., tissue, outside paraffin blocks or slides), blood, serum, plasma, and urine; to be collected after subjects have met eligibility and signed consent. Clinically-indicated samples (e.g., bone marrow, cerebrospinal fluid (CSF), malignant ascites, and effusions) collected under treatment protocols may be transferred to this biorepository protocol for research We will also obtain samples (mainly blood) from volunteer, consenting 1st-3rd degree biological relatives of patients with histologically confirmed cancer, to be paired with their family member.

Tissue will be accessed by study investigators. Additional CCR investigators who wish to use tissue from this repository must first provide a written Letter of Intent, (LOI), to be reviewed by an investigator appointed ad hoc committee for approval.

Assays used for sample processing, establishment of cell lines, patient derived xenograft models, and storage are described in detail within this protocol. Also, some assays for future translational research are either listed or described herein. Further detailed description of experimental designs, along with statistical analysis, will be provided within future investigator-initiated sample use addendums to this protocol, or new IRB approved protocols, developed in order to study samples from this biorepository.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Adult subject (age 18 and older) co-enrolled on a trial, or otherwise undergoing consultation, screening, or follow up on existing protocols conducted at the NIH Clinical Center, who are evaluated in the Women s Malignancies Branch Clinic.
* Participant or biological relative of a participant, as follows:
* Participant with a histologically confirmed breast cancer or other gynecologic malignancy; histopathology of the biopsy tissue must be

confirmed by the NCI Laboratory of Pathology, prior to banking of the tissue on this protocol.

* Biological relative (1st -3rd degree) of a participant who meets the eligibility of histologically confirmed malignancy per above

criterion.

* Subject willingness and ability to provide informed consent.
* Subject willingness to provide tissue samples for banking.

EXCLUSION CRITERIA:

- Pregnant women are not eligible to take part; pregnancy will be assessed using clinical criteria (medical history and physical exam).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are being seen in follow up, consultation, or presenting for enrollment on a clinical trial at the NIH Clinical Center
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-01-04 (Actual); Primary Completion 2028-12-29 (Estimated); Study Completion 2028-12-29 (Estimated)

PRIMARY OUTCOMES:
Establishment of a tissue repository for the collection and banking of tissue samples | at study completion
  A tissue repository

CONTACTS AND LOCATIONS:
Overall Officials: Takeo Fujii, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. @@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2019-C-0025.html